CLINICAL TRIAL: NCT04237194
Title: A New Diagnostic Method to Assess Paclitaxel-Induced Peripheral Neuropathy
Acronym: PacTox
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carsten Dahl Mørch (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Carsten Dahl Mørch, Associate Professor, Aalborg University
Organization: Aalborg University (Other)
Other Study IDs: N-20190071
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Assessment of nerve fiber excitability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the impact of Paclitaxel treatment on the nerve excitability of the small and large nerve fibers

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common side effect of many chemotherapeutic agents, especially antineoplastic agents. To limit the nerve damages, early detection and management of CIPN is crucial and leaves an urgent demand for new diagnostic tools. Perception threshold tracking has enabled assessments of nerve excitability tests of both small and large sensory nerves and may be used to assess CIPN at early stages. The purpose of this study is to examine whether a new nerve excitability test can detect changes in the membrane properties of the small and large nerve fibers during chemotherapy treatment.

In this study nerve excitability tests will be performed with 2 different electrodes using a novel perception threshold tracking technique to assess the Nerve excitability of small and large fibers. Further quantitative sensory tests (QST) will be performed to estimate the vibration threshold, warm and cool perception thresholds, heat and cold pain thresholds, and perceived intensity to static mechanic stimulations will be assessed. Symptoms of CIPN will be assessed using the Common Terminology Criteria for Adverse events scale and a Quality of Life Questionnaire CIPN twenty-item scale.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years
2. Histopathologically verified breast cancer
3. Performance Status according to WHO/ECOG (PS) 0-2
4. Candidate for adjuvant standard treatment with EC and Paclitaxel
5. Not previously treated with chemotherapeutic agents
6. Neurological examination without pathological findings
7. Willingness to voluntarily sign an informed consent

Exclusion Criteria:

1. Previously neoadjuvant treatment with chemotherapy
2. Receives prophylactic bone marrow stimulants
3. HIV
4. Diabetes mellitus
5. Opioid requirement
6. Symptomatic neurosensory disorders
7. Neurological diseases, such as sclerosis and epilepsy
8. Alcohol abuse
9. "Palmar-plantar erythrodysesthesia syndrome" / ulceration of hands or feet
10. Cannot understand written or oral information in Danish
11. Inability to cooperate

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer mainly affects women.
Study Population: Breast cancer patients receiving adjuvant chemotherapy, consisting of 3 cycles of Epirubicin and Cyclophosphamide (EC), followed by 3 cycles of Paclitaxel (9 Paclitaxel infusions).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of Nerve fiber excitability | The difference between baseline and the 6 months follow-up
  The chronaxie and the rheobase to rectangular stimuli, the accommodation to triangular stimuli, and the electrotonus to subthreshold hyperpolarizing pre-pulses for large and small sensory nerves from the excitability measure.

SECONDARY OUTCOMES:
Change of Quantitative sensory test | The difference between baseline and the 6 months follow-up
  The Quantitative sensory test is a reduced version of the German protokol and contains warmth and cold detection thresholds, heat and cold pain thresholds, vibration threshold and perceived intensity to mechanical stimuli.
Changed of CTCAE | The difference between baseline and the 6 months follow-up
  Common Terminology Criteria for Adverse events scale is a scale from 0 to 5, where 5 is worse.
Change of CIPN20. | The difference between baseline and the 6 months follow-up
  Quality of Life Questionnaire Chemotherapy-Induced Peripheral Neuropathy Twenty-Item scale is a 20-item self-report questionnaire. Items are scored 1-4 with 1 representing "not at all" and 4 "very much." Scores are then linearly converted to a 0-100 scale where 100 is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Laurids Ø Poulsen, MD, PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available